CLINICAL TRIAL: NCT01320150
Title: Risk Factors and Mechanisms for Persistent Postsurgical Pain After Total Knee Replacement
Acronym: PPP-TKA
Status: Completed | Type: Observational
Sponsor: Rush University Medical Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Asokumar Buvanendran, Attending Physician, Rush University Medical Center
Other Study IDs: WS735224
Record Dates: First submitted 2011-03-18; First posted 2011-03-22 (Estimated); Results first posted 2019-12-03 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-08

CONDITIONS: Persistent Postsurgical Pain
Keywords: persistent postsurgical pain (PPP)
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA, RNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PPP and Non-PPP: Study Subjects with PPP and without PPP at followup

SUMMARY:
Osteoarthritis (OA) is the single most common cause of disability in mid and late life. About 27 million people in the United States suffer from this incurable process and 10 million have OA of the knee. Total knee replacement (TKR) is a reliable treatment option for patients disabled by knee OA who have failed non-operative treatment; 58% of these surgeries are performed on patients 65 years or older. Despite the overall success of TKR in most cases, persistent postsurgical pain (PPP) of the operated knee remains a common and often difficult to treat postoperative outcome affecting 13-20% of all patients at 6 months post-TKR, which amounts to 65,000-100,000 patients/year in the USA. Important secondary outcomes of PPP are restricted physical mobility and poor quality of life, especially in older patients.

Recent findings spanning the pre-, intra- and postoperative periods suggest that the development of PPP after TKR is a multi-factorial process, comprised of both neurophysiologic and psychosocial factors. Likely determinates include preoperative thermal pain sensitivity, anxiety, pain catastrophizing; and postoperative area of secondary mechanical hyperalgesia or hypoalgesia (numbness). There is already agreement that the intensity of early (acute) postoperative pain is one of the factors predicting PPP. To date, most studies have examined the role of risk factors in isolation and/or within a single domain, and no prospective study has comprehensively evaluated the interaction of neurophysiologic and psychosocial variables in the evolution of PPP following TKR. The lack of information regarding how neurophysiologic pathways and patient cognitive/affective states interact over time following otherwise successful TKR has greatly undermined the understanding of PPP after TKR.

The proposed project is a single-site, prospective study of 300 OA patients aged 18-85 yrs undergoing primary TKR. The study is designed to identify factors from the pre-, intra- and postoperative phases of TKR that contribute to PPP at 6 months. Specific risk factors were selected because they are potentially modifiable, and therefore may be amenable to intervention. Patients will be assessed from pre-surgery to 6 months post surgery. The proposed multi-factorial and prospective approach to investigating risk factors is a vital next step towards understanding the complex phenomenon of PPP.

DETAILED DESCRIPTION:
Overall Strategy: The primary aim of this application is to investigate relationships of risk factors to the development of persistent postoperative pain (PPP) at 6 mo following TKR, through independently predictive and mediated models.

These risk factors are preoperative thermal pain sensitivity, pain anxiety and catastrophizing; postoperative area of secondary mechanical hyperalgesia or hypoalgesia (numbness) and pain intensity. PPP for this study will be defined as "pain in the operated knee at six months after TKR, with other causes of pain excluded and reported intensity on 0-10 Numerical Response Scale (NRS) scale of ≥4". The study will also evaluate the relationship of PPP incidence with the severity of functional impairment. This is a single-site prospective clinical investigation of 300 consented OA patients undergoing primary, unilateral TKR.

ELIGIBILITY:
Inclusion Criteria:

* undergoing standard tricompartmental TKR;
* 18 to 85 yrs of age;
* patient has a diagnosis of osteoarthritis
* knee to be replaced is the primary source of patient's pain;
* patient agrees to preoperative and follow-up visits and to comply with the assessment tests;
* patient consents to standard anesthetic and analgesic protocol, with medical care as deemed necessary by the anesthesiologist, and has no contraindications.

Exclusion Criteria:

* chronic opioid use ≥ 10 mg/day of morphine equivalents within one wk prior to the surgery, and duration of use > 4 wks;
* history of opioid abuse;
* inability to understand and communicate with the investigators to complete the study related questionnaires
* patient currently enrolled in another study;
* patient is planning to undergo another elective joint replacement procedure during the 6-mo period of participation;
* any co-morbidity which results in severe systemic disease limiting function {as defined by the American Society of Anesthesiology (ASA) physical status classification > 3}

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Osteoarthritis patients at the RUSH university medical center undergoing primary, unilateral TKR
Sampling Method: Probability Sample
Enrollment: 311 (Actual)
Dates: Start 2011-03; Primary Completion 2017-08 (Actual); Study Completion 2018-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Asokumar Buvanendran, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Result] Buvanendran A, Della Valle CJ, Kroin JS, Shah M, Moric M, Tuman KJ, McCarthy RJ. Acute postoperative pain is an independent predictor of chronic postsurgical pain following total knee arthroplasty at 6 months: a prospective cohort study. Reg Anesth Pain Med. 2019 Mar;44(3):e100036. doi: 10.1136/rapm-2018-100036. Epub 2019 Feb 15. PMID 30770420

RESULTS

PARTICIPANT FLOW:
Groups:
- All Study Participants: Study Subjects with and without Persistent Post-operative Pain (PPP) at followup
Period: Overall Study
Arm/Group | All Study Participants
Started | 311
PPP (Subjects with Persistent Post-Operative Pain (PPP)) | 34
Non-PPP (Subjects without Persistent Post-Operative Pain (Non-PPP)) | 211
Completed | 245
Not Completed | 66
Not completed — Protocol Violation | 15
Not completed — Withdrawal by Subject | 5
Not completed — Death | 2
Not completed — Lost to Follow-up | 44

BASELINE CHARACTERISTICS:
Population: Persistent Post-surgical Pain (PPP) and Non-PPP groups are defined at 6 month follow-up.
Groups:
- Non PPP: Those without Persistent Post-surgical Pain (PPP)
- Persistent Post Surgical Pain (PPP): Those with Persistent Post-surgical Pain (PPP)
- Total: Total of all reporting groups
Arm/Group | Non PPP | Persistent Post Surgical Pain (PPP) | Total
Number analyzed (Participants) | 211 | 34 | 245
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 65 [61 to 70] | 64 [53 to 69] | 65 [60 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 133 | 27 | 160
  Male | 78 | 7 | 85
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 159 | 20 | 179
  African American | 52 | 14 | 66

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Post-Operative Persistent Pain (PPP)
Description: PPP for this study will be defined as "pain in the operated knee at six months after Total Knee Replacement surgery, with other causes of pain excluded, and a reported intensity on 0-10 Numerical Response Scale (NRS) of ≥4 where higher pain scores indicate higher levels of pain. NRS scores range from 0 {No Pain} to 10 {Worst Imaginable Pain}.
Time Frame: 6 months postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | PPP and Non-PPP
Number analyzed (Participants) | 245
Participants
  non PPP | 211
  PPP | 34

ADVERSE EVENTS:
Time Frame: Subjects were followed for 6 months
Description: Subject were identified by group (PPP, non-PPP) at the end of the 6 month follow-up, so adverse events is based on one unified group.
Arm/Group | All Study Participants
All-Cause Mortality (participants affected / at risk) | 2/311
Serious Adverse Events (participants affected / at risk) | 0/311
Other Adverse Events (participants affected / at risk) | 0/311

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-01): https://cdn.clinicaltrials.gov/large-docs/50/NCT01320150/Prot_SAP_000.pdf